CLINICAL TRIAL: NCT07300579
Title: Vascular Events in Noncardiac Surgery Patients Cohort Evaluation Study 2
Acronym: VISION-2
Status: Not yet recruiting | Type: Observational
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Population Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 1.0.2025.08.25
Record Dates: First submitted 2025-12-10; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: Myocardial Injury After Noncardiac Surgery (MINS); Bleeding Independently Associated With Mortality After Noncardiac Surgery (BIMS); Sepsis; Infection Without Sepsis; Post-operative Complications
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Continuous vital signs measurement device — In this observational study, enrolled participants will wear the Vitaliti™ CVSM-1A device continuously before surgery, wherever and whenever possible, or as soon as possible after surgery and for up to 30-days after surgery. We will collect continuous biometric data using the Vitaliti™ CVSM-1A device. Patients, healthcare providers, data collectors, and outcome adjudicators will be blind to the Vitaliti™ data. Data from participants will be analyzed to determine the pattern and frequency of physiological precursors to outcome events. This data will be used to inform machine learning algorithms for prediction and early detection of post-surgical complications. A biobank will also be established to support exploratory proteomic and genotyping analyses to better understand biological mechanisms underlying post-operative complications.

SUMMARY:
VISION-2 is an international, multi-site, prospective observational cohort study of 20,000 patients undergoing noncardiac surgery. Continuous biometric data will be blindly collected for the first 30 postoperative days, in hospital and at home, using Vitaliti™. Following study enrollment and baseline data collection, follow up visits will occur in-hospital, at 30-days, and 1-year post-operatively.

VISION-2 has 3 primary objectives, among participants who underwent noncardiac surgery, we will: 1) determine the pattern and frequency of physiological precursors (i.e., biophysical signals) to MINS, BIMS, sepsis, and infection without sepsis; 2) build prediction models from these biophysical signals and their extracted features through supervised machine learning, for the prediction and early detection of those complications; and 3) build a biobank for evaluation of novel biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥65 years;
2. underwent non-cardiac surgery with general, neuraxial, local, or regional anesthesia; and
3. expected to require an overnight hospital admission after surgery.

Exclusion Criteria:

1. hearing aid(s) or cochlear implant(s) in left ear;
2. pacemaker/implantable cardioverter-defibrillator (ICD);
3. externally programmable cerebrospinal fluid shunt;
4. deep brain stimulator;
5. intolerance/allergy to adhesive;
6. history of dementia, or;
7. previous enrollment in the VISION-2 Study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients 65 years of age and older undergoing non-cardiac surgery with anesthesia expected to require an overnight hospital admission
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2030-02 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Myocardial injury after noncardiac surgery (MINS) | 30 days after surgery
  MINS not meeting 4th definition of MI is an elevated troponin measurement that occurs during the first 30 days after surgery that is judged as resulting from myocardial ischemia AND does not fulfill the MI definition. The following defines elevated troponin measurement for the diagnosis of MINS during the first 30 days after surgery: non high sensitivity Troponin T assay: ≥0.03 µg/L; high sensitivity Troponin T assay: between 20 - <65 ng/L with an absolute change ≥5 ng/L or a value ≥65 ng/L; DVIA Centaur Siemens high-sensitivity cardiac troponin I: ≥75 ng/L; ARCHITECT STAT Abbott Laboratories high-sensitivity cardiac troponin I ≥60 ng/L; other troponin assays: any measurement above the 99th percentile of the upper reference limit.
Bleeding independently associated with mortality after noncardiac surgery (BIMS) | 30 days after surgery
  A bleeding meeting any of the following 3 criteria: a) leading to a postoperative hemoglobin <70 g/L; b) requiring transfusion of one or more units of red blood cells; c) judged to be the immediate cause of death
Sepsis | 30 days after surgery
  Based on the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3) criteria, sepsis will require a quick Sequential Organ Failure Assessment (qSOFA) Score ≥2 points due to infection. The qSOFA includes the following items and scoring system: a) Glasgow Coma Scale (GCS) score of 13 or less (1 point); b) systolic blood pressure of 100 mm Hg or less (1 point); and c) respiratory rate of 22 breaths/min or more (1 point).
Infection without sepsis | 30 days after surgery
  Pathologic process caused by the invasion of normally sterile tissue or fluid or body cavity by pathogenic or potentially pathogenic organisms.
All-cause mortality | 30 days after surgery
  Death by any cause

SECONDARY OUTCOMES:
Vascular mortality | 30 days and 1 year after surgery
  Any death with a vascular cause and includes those deaths following a myocardial infarction, cardiac arrest, stroke, cardiac revascularization procedure (i.e., percutaneous coronary intervention [PCI] or coronary artery bypass graft [CABG] surgery), heart failure, pulmonary embolus, cardiovascular hemorrhage (i.e., hemorrhage causing cardiac tamponade, non-traumatic vascular rupture [e.g., aortic aneurism, cerebrovascular aneurism], non-stroke intracranial hemorrhage), or deaths due to an unknown cause.
Myocardial infarction (MI) | 30 days and 1 year after surgery
  The definition of myocardial infarction follows the 4th universal definition
Stroke | 30 says and 1 year after surgery
  An acute episode of neurological dysfunction consistent with an ischemic or hemorrhagic cause. For the diagnosis of stroke, the following criteria must be fulfilled: a) rapid onset of a focal/global neurologic deficit with at least one of the following: change in level of consciousness, hemiplegia, hemiparesis, numbness or sensory loss affecting one side of the body, dysphagia/aphasia, hemianopia, amaurosis, or other new neurological signs/symptoms consistent with stroke; b) the duration of a focal/global neurologic deficit is at least 24 hours, OR the neurological deficit results in death, OR there is neuroimaging evidence of a new infarct/ hemorrhage; and c) there is no other readily identifiable non-stroke cause for the clinical presentation (e.g., brain tumor, trauma, infection, hypoglycemia, peripheral lesion).
Proximal venous thromboembolism (VTE) | 30 days and 1 year after surgery
  Proximal VTE includes pulmonary embolism or proximal deep vein thrombosis.
Proximal deep venous thrombosis (DVT) | 30 days and 1 year after surgery
  The diagnosis of proximal deep venous thrombosis requires:
  Thrombosis involving the popliteal vein or more proximal veins for leg DVT or axillary or more proximal veins for arm DVTs.
  Any of the following defines evidence of vein thrombosis:
  A persistent intraluminal filling defect on contrast venography (including on computed tomography), Noncompressibility of one or more venous segments on B mode compression ultrasonography, or a clearly defined intraluminal filling defect on doppler imaging in a vein that cannot have compressibility assessed (e.g., iliac, inferior vena cava, subclavian).
Pulmonary embolism (PE) | 30 days and 1 year after surgery
  The diagnosis requires symptoms and any one of the following:
  1. a high probability ventilation/perfusion lung scan,
  2. an intraluminal filling defect of segmental or larger artery on a helical CT scan,
  3. an intraluminal filling defect on pulmonary angiography, or
  4. a positive diagnostic test for DVT (e.g., positive compression ultrasound) and one of the following:
  i) non-diagnostic (i.e., low or intermediate probability) ventilation/perfusion lung scan, or ii) non-diagnostic (i.e., subsegmental defects or technically inadequate study) helical CT scan
Acute kidney injury (AKI) | 30 days and 1 year after surgery
  Increase in serum creatinine concentration from the preoperative (pre-enrollment) concentration by either an increase of ≥26.5 μmol/L (≥0.3 mg/dL) within 48 hours of surgery or an increase of 50% or greater within 7 days of surgery.
New acute renal failure resulting in dialysis | 30 days and 1 year after surgery
  New acute renal failure resulting in use of a hemodialysis machine or peritoneal dialysis apparatus
Acute heart failure | 30 days and 1 year after surgery
  Acute Heart Failure is defined as a clinical sign (i.e., at least one of the following: elevated jugular venous pressure, respiratory rales/crackles, crepitations, or presence of S3) and at least one of the following:
  1. Radiographic findings (i.e., at least one of the following: vascular redistribution, interstitial pulmonary edema, frank alveolar pulmonary edema, or multiple and diffuse bilateral B lines on ultrasonography);
  2. Elevated levels of natriuretic peptides; or
  3. Heart failure treatment implemented with diuretics with documented clinical improvement.
New clinically important atrial fibrillation | 30 days and 1 year after surgery
  The definition of clinically important atrial fibrillation requires the documentation of atrial fibrillation of any duration on an ECG or rhythm strip, which results in angina, congestive heart failure, symptomatic hypotension, or requires treatment with a rate controlling drug, antiarrhythmic drug, or electrical cardioversion.
Nonfatal cardiac arrest | 30 days and 1 year after surgery
  Successful resuscitation from either documented or presumed ventricular fibrillation, sustained ventricular tachycardia, asystole, or pulseless electrical activity requiring cardiopulmonary resuscitation, pharmacological therapy, or cardiac defibrillation.
Life-threatening bleeding | 30 days and 1 year after surgery
  Life-threatening bleeding is bleeding that is fatal or leads to: significant hypotension that requires inotrope or vasopressor therapy, or urgent (within 24 hours) surgery (other than superficial vascular repair).
Critical organ bleeding | 30 days and 1 year after surgery
  A critical organ bleeding event is bleeding that was intracranial, intraocular, intraspinal, pericardial, retroperitoneal, or intramuscular with compartment syndrome.
Peripheral arterial thrombosis | 30 days and 1 year after surgery
  We will consider a peripheral arterial thrombosis to have occurred where there is clear evidence of abrupt occlusion of a peripheral artery (i.e., not a stroke, myocardial infarction, or pulmonary embolism) consistent with either an acute local thrombotic event or a peripheral arterial embolism. To fulfill this definition, we require at least one of the following objective findings of peripheral arterial thrombosis:
  1. Surgical report indicating evidence of arterial thrombosis/ peripheral arterial embolism;
  2. Pathological specimen demonstrating arterial thrombosis/ peripheral arterial embolism;
  3. Imaging evidence consistent with arterial thrombosis/ peripheral arterial embolism; or
  4. Autopsy reports documenting arterial thrombosis/ peripheral arterial embolism
Amputation | 30 days and 1 year after surgery
  Any amputation procedure, or auto amputation after the initial surgery.
Delirium | 30 days and 1 year after surgery
  For the diagnosis of delirium any one of the following criteria is required:
  1. Patient meets the criteria for delirium on any in-person delirium assessment based on the Confusion Assessment Method (CAM) or any of its operationalizations (e.g., 3D-CAM, CAM-ICU); OR
  2. Positive history of delirium based on the review of hospital health records.
Pneumonia | 30 days and 1 year after surgery
  An acute infection of the pulmonary parenchyma that is associated with at least one sign or symptom of lower respiratory acute infection (e.g., cough, pleuritic chest pain) or acute systemic illness (e.g., fever, chills, confusion, hypoxemia); accompanied by the presence of an acute infiltrate/consolidation on a chest radiograph or auscultatory findings consistent with pneumonia (such as crackles and/or localized rales) for which there is no other explanation.
Surgical site infection | 30 days and 1 year after surgery
  An infection that involves the skin, subcutaneous tissue of the incision (superficial incisional), or the deep soft tissue (e.g., fascia, muscle) of the incision (deep incisional).
Urinary tract infection | 30 days and 1 year after surgery
  An infection that involves the urinary tract.
Clinically important ileus | 30 days and 1 year after surgery
  Physician diagnosis of functional obstruction of the gastrointestinal tract in the absence of an alternative diagnosis that leads to postoperative decreased bowel activity. The definition requires the following criteria:
  1. inability to pass flatus or stool for >24 hours; and
  2. persistence of one or more of the following signs and symptoms for >24h (abdominal distention; diffuse abdominal pain; or nausea or vomiting.
Falls | 30 days and 1 year after surgery
  Fall from standing height or walking
Post-discharge acute hospital care | 30 days after surgery
  A composite outcome of hospital re-admission and emergency department visit, which includes urgent-care centre visit.
Emergency department visit | 30 days after surgery
  Visit to an emergency department, which includes urgent-care centre visits.
Rehospitalization | 30 days after surgery
  Admission to acute care hospital after initial discharge from hospital for index surgery.
Sepsis | 1 year after surgery
  The Third International Consensus Definitions Task Force defines sepsis as a "life-threatening organ dysfunction due to a dysregulated host response to infection." Based on the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3) criteria, sepsis will require a quick Sequential Organ Failure Assessment (qSOFA) Score ≥2 points due to infection. The qSOFA includes the following items and scoring system:
  1. Glasgow Coma Scale (GCS) score of 13 or less (1 point),
  2. systolic blood pressure of 100 mm Hg or less (1 point), and
  3. respiratory rate of 22 breaths/min or more (1 point).
Infection without sepsis | 1 year after surgery
  Pathologic process caused by the invasion of normally sterile tissue or fluid or body cavity by pathogenic or potentially pathogenic organisms.

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Hamilton General Hospital, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Juravinski Hospital & Cancer Centre, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No